CLINICAL TRIAL: NCT04163250
Title: Prognostic Value of Urinary TIMP-2/ IGFBP7 in Intra-Arterial Contrast-Associated Acute Kidney Injury
Brief Title: Use of Urinary Cell-Cycle Arrest Biomarkers in Contrast-Associated Nephropathy After Coronary Angiography
Status: Completed | Type: Observational
Sponsor: Eva de Miguel Balsa (Other)
Responsible Party: Sponsor-Investigator, Eva de Miguel Balsa, Principal Investigator, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Organization: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Other Study IDs: GV/2019/003
Record Dates: First submitted 2019-11-10; First posted 2019-11-14 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Contrast-induced Nephropathy
Keywords: Contrast media; Urinary cell-cycle arrest biomarkers; Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with ACS undergoing cardiac catheterization: Adults with moderate / high risk acute coronary syndrome undergoing coronary intervention.
  The sample will be selected consecutively, including patients admitted to the Cardiac Coronary Unit and who require a radiological test with intra-arterial IC administration, for diagnostic or diagnostic / therapeutic purposes
  Interventions: Diagnostic Test: Urinary determination of TIMP-2/ IGFBP7

INTERVENTIONS:
Diagnostic Test: Urinary determination of TIMP-2/ IGFBP7 — Urinary determination of TIMP2-IGFBP7 in the an urine sample obtained within 12 hours prior to contrast administration. A single determination will be made, which will be sent to the laboratory. The doctor who treats the patient will not know the result of the test, and the treatment will not be influenced by the result.
  According to the manufacturer, 10 ml of fresh urine should be collected in a sterile container and the laboratory should centrifuge them within the time of collection.
  The result is reported as a single value calculated as the concentration of TIMP-2 (ng / mL) multiplied by the concentration of IGFBP7 (ng / mL) divided by 1000. The result is reported without units.

SUMMARY:
Radiological examinations that require the administration of iodinated contrasts (IC) for diagnostic and therapeutic purposes are essential in current clinical practice, and their use in interventional procedures has been progressively increasing.

IC can cause kidney damage, so there is caution in their use in at-risk populations. This fact may limit its diagnostic use, with data on underutilization of interventional techniques in patients with renal insufficiency, which worsen their prognosis.

In addition, once the use of IC contrasts is decided, preventive measures, such as hyperhydration,are used and can have potential side effects, especially in patients at risk of heart failure (acute coronary syndrome, low left ventricular ejection fraction).

New biomarkers of kidney damage have recently been developed, based on the detection of molecules expressed by the kidney in situations of early damage. The quantitative determination of cell cycle arrest proteins (Tissue Inhibitor of metalloproteinase 2 (TIMP2) and Insulin-Like Growth Factor Binding Protein -7 (IGFBP7)) can be predictive of the development of moderate to severe contrast-associated acute kidney injury.

Urinary determination of [TIMP-2] x [IGFBP7] in patients with ACS (acute coronary syndromes) before cardiac catheterization would allow early identification of those patients vulnerable to IC-induced toxicity and adjustment of preventive measures.

DETAILED DESCRIPTION:
Urinary determination of [TIMP-2] x [IGFBP7] in patients with ACS undergoing cardiac catheterization would allow early identification of those patients vulnerable to IC-induced toxicity and adjustment of both appropriate preventive measures.

A prospective, descriptive observational study will be carried out to determine sensitivity and specificity of the urinary determination of TIMP2-IGFBP7 and predictive values in the early diagnosis of contrast-associated acute kidney injury (AKI) in patients admitted to the Coronary Care Unit (CCU) in a spanish hospital.

OBJECTIVES

* PRIMARY OBJECTIVE: To determine the operational characteristics (sensitivity, specificity) of the TIMP2-IGFBP7 biomarker in routine clinical practice, in the early diagnosis of contrast-induced AKI (acute renal injury) in patients admitted to the CCU, exposed to iodinated contrasts. The established renal failure is defined as KDIGO (Kidney Disease Improving Global Outcomes) stage ≥ 2 in the 24 to 72 hours after the administration of contrasts.
* SECONDARY OBJECTIVES

Evaluate these parameters according to the patient's initial risk level:

* Estimated renal function upon admission
* Initial severity estimated by GRACE score
* Sex
* Age
* Contrast media type and volume
* Patient weight
* Dose of contrast
* Diabetes

A single determination (10 ml of fresh urine) should be collected in a sterile container and the laboratory should centrifuge them within the time of collection. Neither the attending physicians nor the investigators will know the results, and the treatment will not be influenced.

The result is reported as a single value which is the concentration of TIMP-2 (ng / mL) multiplied by the concentration of IGFBP7 (ng / mL) divided by 1000. The result is reported without any unit or concentrations of individual biomarkers. As previously reported, a value of> 0.3 identifies patients with a high probability of presenting a moderate to severe AKI (acute kidney injury) in 12 hours, while a value of ≤ 0.3 identifies patients with a low risk of developing a moderate to serious AKI

An aliquot of urine will be stored at -80 ° C in the Clinical Analysis Department

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 21 years exposed to intra-arterial iodinated contrast media for diagnostic / therapeutic purposes and who have signed the Informed Consent document.

Exclusion Criteria:

* Patients who have been exposed to a previous dose of iodinated contrast within 72 hours prior to recruitment.
* Patients with urgent radiodiagnostic intervention criteria, when it is not possible to obtain a previous urine sample without delaying the diagnosis and / or the intervention.
* Patients in anuria.
* Patients with chronic kidney disease, treated with hemodialysis (HD) or peritoneal dialysis.
* Bilirubinuria: bilirubin concentrations in the urine> 7.2 g / dL interfere with the result.
* Patients in terminal situations, in which diagnostic and therapeutic tests are limited.
* Patients under 21 years.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 21 years, with moderate / high risk acute coronary syndrome according to GRACE score and exposed to intra-arterial iodinated contrast media
Sampling Method: Non-Probability Sample
Enrollment: 194 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Contrast-Associated Acute Kidney Injury | up to 72 hours of exposure
  Absolute increase of 0.3 mg / dl in the creatinine value and / or a relative increase greater than 1.5 times the baseline creatinine value, measured at 48 and 72 hours after exposure to contrast.

SECONDARY OUTCOMES:
Mortality | up to 30 days
  Patients who die during their hospital stay for any reason
Need of renal replacement techniques | From exposure to contrasts to three months
  Hemodialysis, peritoneal dialysis or continuous renal replacement techniques,

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General Universitario de Elche, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: Undecided